CLINICAL TRIAL: NCT04544267
Title: Efficacy, Immunogenicity, and Safety of High-Dose Quadrivalent Influenza Vaccine Compared With Standard-Dose Quadrivalent Influenza Vaccine in Children 6 Months Through 35 Months of Age
Brief Title: Study on a High-Dose Quadrivalent Influenza Vaccine Compared With Standard-Dose Quadrivalent Influenza Vaccine in Children 6 Months Through 35 Months of Age
Acronym: QHD00014
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was interrupted due to COVID-19 pandemic and terminated due to new changes to the recommendations for flu vaccines
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD00014; U1111-1243-5993 (Registry Identifier: ICTRP); QHD00014 (Other: Sanofi Identifier); 2019-004721-24 (EudraCT Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: A sentinel safety cohort was selected for collection safety events where QIV-HD was administered open-label in 100 participants. These subjects did not provide blood samples and were not followed for influenza-like illness (ILI) surveillance.
  A re-vaccination cohort was composed of a subset of approximately 120 participants from Season 1 (2021-2022 Northern Hemisphere) were re-enrolled and re-randomized in Season 3. The re-vaccination cohort was included, re-randomized to receive either QIV-HD or QIV-SD, provided blood samples in Season 1 and Season 3, and were not followed for ILI surveillance during their participation in Season 3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A total of 100 participants were in an uncontrolled, open-label sentinel cohort, while all other participants were in an randomized, modified double-blind design. The following measures ensured the integrity of the blinded data for the participants in the randomized, modified double-blind cohort:
  * The unblinded qualified study staff member, independent of the safety evaluation and other study evaluations, administered the vaccine
  * The Investigators (or delegates) in charge of safety assessment, the study staff who collect the safety data, and the laboratory personnel who analyze the blood samples did not know which product was administered
  * The participant / parent / guardian did not know which product was administered. To maintain the blinding of the participant / parent / guardian, the vaccine syringe label was covered with appropriate materials prior to administration.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QIV-HD (Experimental): One injection of QIV-HD on Day 0. For participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered on Day 28.
  Interventions: Biological: Quadrivalent influenza vaccine, high-dose
- QIV-SD (Active Comparator): One injection of QIV-SD on Day 0. For participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered on Day 28.
  Interventions: Biological: Quadrivalent influenza vaccine, standard dose

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine, high-dose — Pharmaceutical form: suspension for injection in a pre-filled syringe; route of administration: intramuscular
  Arms: QIV-HD
Biological: Quadrivalent influenza vaccine, standard dose — Pharmaceutical form: suspension for injection in a pre-filled syringe; route of administration: intramuscular
  Arms: QIV-SD

SUMMARY:
The primary objective of the study was to compare the clinical efficacy of high-dose quadrivalent influenza vaccine (QIV-HD) to standard-dose quadrivalent influenza vaccine (QIV-SD) in participants 6 months through 35 months of age for the prevention of laboratory-confirmed influenza illness caused by any influenza A or B type.

The secondary objectives of the study were:

* To compare QIV-HD to QIV-SD:
* in participants 6 months through 35 months of age for the prevention of laboratory-confirmed influenza illness caused by any influenza A or B type using a more stringent threshold
* in participants 6 months through 35 months of age for the prevention of laboratory-confirmed protocol-defined influenza-like illness caused by viral strains similar to those contained in the vaccine.
* in participants 6 months through 23 months of age for the prevention of laboratory-confirmed influenza illness caused by any influenza A or B types.
* To compare hemagglutination inhibition (HAI) immune response of QIV-HD to QIV-SD in participants 6 months through 35 months of age
* To describe the HAI, seroneutralization (SN), and anti-neuraminidase (NA) immune response
* To describe the immune response to revaccination in Season 3 (Northern Hemisphere)
* To describe the safety profile of each vaccine

DETAILED DESCRIPTION:
The study was planned to start in the second half of 2020 with the Sentinel Safety Cohort. Following the Sentinel Safety Cohort, the main efficacy cohort was to be conducted during the 2021-2022 Northern Hemisphere influenza season (Season 1), the 2021-2022 Southern Hemisphere influenza season (Season 2), and the 2021-2022-2023 Northern Hemisphere influenza season (Season 3).

Participants received either 1 or 2 doses of the study vaccine depending on whether they were previously influenza vaccinated or previously influenza unvaccinated, respectively.

Study duration per participant was approximately 6 to 7 months.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 to 35 months on the day of the first study visit
* Informed consent form was signed and dated by the parent(s) or guardian(s) and by an independent witness, if required by local regulations.
* Participant and parent / guardian who were able to attend all scheduled visits and to comply with all study procedures.
* Covered by health insurance if required by local regulations
* For Season 3 Re-vaccination Cohort: eligible participants must have been enrolled in the Season 1 (2021-2022 Northern Hemisphere season) immunogenicity subset and must have completed all study procedures (ie, blood draws and vaccinations) in Season 1.

Exclusion criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* For all participants: Receipt of any vaccine in the 30 days preceding the first study vaccination. For participants in immunogenicity subset: Planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza in the preceding 6 months with either the study vaccine or another influenza vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency (eg, HIV); or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances. Exception: participants with an egg allergy are allowed to enroll in the study.
* Thrombocytopenia, bleeding disorder, or receipt of anticoagulants that based on Investigator's judgment contraindicate intramuscular vaccination
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C [≥ 100.4 F]). A prospective participant would not be included in the study until the condition was resolved or the febrile event was subsided.
* Identified as natural or adopted child of the Investigator or employee with direct involvement in the proposed study.
* Personal or family history of Guillain-Barre Syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant development delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* For Season 3 (2022-2023 Northern Hemisphere) main cohort: participants who were enrolled in a previous study season are excluded from Season 3, with the exception of the Re-vaccination Cohort.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (10):
- United States (10):
  - California Research Foundation Site Number : 8400008, San Diego, California
  - Acevedo Clinical Research Associates Site Number : 8400007, Miami, Florida
  - Emory Childrens Center- Site Number : 8400001, Atlanta, Georgia
  - Heartland El Dorado- Site Number : 8400032, El Dorado, Kansas
  - Kentucky Pediatrics / Adult Research- Site Number : 8400005, Bardstown, Kentucky
  - Velocity Clinical Research- New Orleans Site Number : 8400009, New Orleans, Louisiana
  - Ohio Pediatric Research- Site Number : 8400027, Dayton, Ohio
  - Rainbow Pediatrics- Site Number : 8400033, Barnwell, South Carolina
  - Cenexel JBR- Site Number : 8400006, Salt Lake City, Utah
  - Foothill Family Clinic South- Site Number : 8400045, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: QHD00014 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25341&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sentinel safety cohort of the study was conducted at 10 centers from 15 September 2020 to 10 May 2021.
Pre-assignment Details: The sentinel safety cohort of 100 participants were enrolled in the study. This study was prematurely terminated following a global shift in the influenza vaccine composition from quadrivalent to trivalent formulation for 2024-2025 season. Hence, main efficacy cohort was not conducted, and the safety analysis of the sentinel cohort was presented.
Groups:
- Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose: Participants who were previously vaccinated against influenza received 1 dose of quadrivalent influenza vaccine (split virion, inactivated) high-dose (QIV-HD) intramuscular (IM) injection on Day 0.
  Participants who were not previously vaccinated against influenza received 1 dose of QIV-HD IM injection on Day 0 and 1 dose on Day 28.
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Expanded safety analysis set included participants who received at least 1 dose of the study vaccine in the sentinel safety cohort.
Groups:
- Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose: Participants who were previously vaccinated against influenza received 1 dose of QIV-HD IM injection on Day 0.
  Participants who were not previously vaccinated against influenza received 1 dose of QIV-HD IM injection on Day 0 and 1 dose on Day 28.
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.7 (0.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 20
  White | 71
  Mixed Origin | 6
  Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laboratory-Confirmed Influenza Illness Caused by Any Influenza Viral Types/Subtypes
Description: Laboratory-confirmed influenza was a positive influenza result on either polymerase chain reaction (PCR) or viral culture. An influenza-like illness (ILI) was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches).
Time Frame: From 14 days after the first vaccine administration up to 6 months after the last vaccine administration (vaccines administered at Days 0 and 28), approximately 196 days
Population: The main efficacy cohort was not conducted due to shift in the global influenza vaccine guidelines. Hence, no analysis was performed.
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine
Description: Laboratory-confirmed influenza was a positive influenza result on either PCR or viral culture. An ILI was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches).
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive in Participants Aged 6 Through 23 Months for Any Influenza A or B Type
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Any Influenza A or B Type According to Previous Vaccination Status
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine According to Previous Vaccination Status
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Any Influenza A or B Type and Associated With Acute Otitis Media (AOM)
Description: Laboratory-confirmed influenza was a positive influenza result on either PCR or viral culture. An ILI was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches). The AOM was based on clinical diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine and Associated With Acute Otitis Media
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Any Influenza A or B Type and Associated With Acute Lower Respiratory Infection (ALRI)
Description: Laboratory-confirmed influenza was a positive influenza result on either PCR or viral culture. An ILI was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches). The ALRI was based on a clinical and/or x-ray diagnosis.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine and Associated With Acute Lower Respiratory Infection
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Influenza-Like Illness Polymerase Chain Reaction-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine
Description: The PCR-confirmed influenza was a positive influenza result on PCR. An ILI was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches).
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Influenza-Like Illness Culture-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine
Description: Culture-confirmed influenza was a positive influenza result on viral culture. An ILI was occurrence of fever concurrently with at least 1 of the following symptoms: cough, wheezing, difficulty breathing, nasal congestion, rhinorrhea, pharyngitis (sore throat), otitis, vomiting, diarrhea, shivering (chills), fatigue (tiredness), headache, or myalgia (muscle aches).
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Influenza-Like Illness Polymerase Chain Reaction-Confirmed as Positive for Any Influenza A or B Types
Description: as for outcome 10
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Influenza-Like Illness Culture-Confirmed as Positive for Any Influenza A or B Types
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Any Influenza A or B Types and Associated With Hospitalization
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Influenza-Like Illness Laboratory-Confirmed as Positive for Viral Strains Similar to Those Contained in the Vaccine and Associated With Hospitalization
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

16. Secondary Outcome: Geometric Mean Titer of Influenza Vaccine Antibodies
Description: Antibody titers were measured by hemagglutination inhibition (HAI) assay.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With Seroconversion
Description: Seroconversion for participants with a pre-vaccination titer <10 [1/dilution (dil)]: Post-injection titer >=40 (1/dil) on 28 days after the last vaccination or significant increase. Seroconversion for participants with a pre-vaccination titer >=10 (1/dil): >=4-fold increase from pre- to post-injection titer on 28 days after the last vaccination. Antibody titers were measured by HAI assay.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Influenza Vaccine Antibody Titer >=10 (1/Dilution)
Description: Antibody titers were measured by HAI assay. The influenza vaccine antibody titer level assessed was >=10 (1/dil).
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

19. Secondary Outcome: Influenza Vaccine Antibody Titer Ratio
Description: Antibody titer ratio was calculated as individual antibody titer 28 days after the last vaccination (Day 56) divided by individual antibody titer at Day 0. Antibody titers were measured by HAI assay.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

20. Secondary Outcome: Number of Participants With Influenza Vaccine Antibody Titer >=40 (1/Dilution)
Description: Antibody titers were measured by HAI assay. The influenza vaccine antibody titer level assessed was >=40 (1/dil).
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

21. Secondary Outcome: Influenza Seroneutralization (SN) Antibody Titer
Description: The antibody titers were measured by the SN method.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

22. Secondary Outcome: Influenza Seroneutralization Antibody Titer Ratio
Description: Antibody titer ratio was calculated as fold increase in serum SN post-vaccination relative to Day 0. Antibody titers were measured by the SN method.
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Participants With Influenza Seroneutralization Antibody Titer >=20 (1/Dilution), >=40 (1/Dilution) and >=80 (1/Dilution)
Description: Antibody titers were measured by the SN method. The SN antibody titer levels assessed were >=20 (1/dil), >=40 (1/dil) and >=80 (1/dil).
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

24. Secondary Outcome: Number of Participants With Influenza Seroneutralization Antibody Titer >=2 and >=4 Fold-Rise
Description: Increase of titer levels >=2 and >=4 were assessed. Antibody titers were measured by the SN method.
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

25. Secondary Outcome: Detectable Influenza Seroneutralization Antibody Titer
Description: Detectable antibody titers were >=10 (1/dil). Antibody titers were measured by the SN method.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

26. Secondary Outcome: Anti-Neuraminidase (Anti-NA) Antibody Titer
Description: Antibody titers were measured by enzyme-linked lectin assay.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

27. Secondary Outcome: Anti-Neuraminidase Antibody Titer Ratio
Description: Antibody titer ratio was calculated as fold increase in anti-NA antibodies post-vaccination relative to Day 0. Antibody titers were measured by enzyme-linked lectin assay.
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

28. Secondary Outcome: Number of Participants With Anti-Neuraminidase Antibody Titer >=20 (1/Dilution), >=40 (1/Dilution) and >=80 (1/Dilution)
Description: Antibody titers were measured by enzyme-linked lectin assay. Anti-NA antibody titer levels assessed were >=20 (1/dil), >=40 (1/dil) and >=80 (1/dil).
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

29. Secondary Outcome: Number of Participants With Anti-Neuraminidase Antibody Titer >=2 and >=4 Fold-Rise
Description: Increase of titer levels >=2 and >=4 were assessed. Antibody titers were measured by enzyme-linked lectin assay.
Time Frame: Day 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

30. Secondary Outcome: Detectable Anti-Neuraminidase Antibody Titer
Description: Detectable antibody titers were >=10 (1/dil). Antibody titers were measured by enzyme-linked lectin assay.
Time Frame: Days 0 and 56
Population: as for outcome 1
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 0

31. Secondary Outcome: Number of Participants With Unsolicited Systemic Adverse Events (AEs) After Each Vaccine Dose Administration
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. Immediate events were recorded to capture medically relevant unsolicited systemic AEs which occurred within the first 30 minutes after vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, pre-listed in the case report form in terms of diagnosis and onset window post-vaccination.
Time Frame: Within 30 minutes after each vaccine administration (vaccines administered at Days 0 and 28)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Participants | 0

32. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions After Each Vaccine Dose Administration
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and case report form, and were considered to be related to the study vaccine administered. An injection site reaction was an AR at and around the injection site of the study vaccine.
Time Frame: Within 7 days after each vaccine administration (vaccines administered at Days 0 and 28)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Participants | 51

33. Secondary Outcome: Number of Participants With Solicited Systemic Reactions After Each Vaccine Dose Administration
Description: A solicited reaction was an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and case report form, and were considered to be related to the study vaccine administered. Systemic AR were all ARs that were not injection site reactions.
Time Frame: Within 7 days after each vaccine administration (vaccines administered at Days 0 and 28)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Participants | 46

34. Secondary Outcome: Number of Participants With Unsolicited Adverse Events After Each Vaccine Dose Administration
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, pre-listed in the case report form in terms of diagnosis and onset window post-vaccination.
Time Frame: Within 28 days after each vaccine administration (vaccines administered at Days 0 and 28)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Participants | 25

35. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was 1 of scientific and medical concern specific to the Sponsor's study vaccine or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor could be appropriate.
Time Frame: From first dose of study vaccine administration (Day 1) up to 6 months after the last vaccine administration (vaccines administered at Days 0 and 28), approximately 210 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
Number analyzed (Participants) | 100
Participants
  SAE | 1
  AESI | 0

ADVERSE EVENTS:
Time Frame: From first dose of study vaccine administration (Day 1) up to 6 months after the last vaccine administration (vaccines administered at Days 0 and 28), approximately 210 days.
Description: Analysis was performed on the expanded safety analysis set.
Arm/Group | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 65/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose (N=100)
Otitis Media Acute (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine (Split Virion, Inactivated) High-Dose (N=100)
Decreased Appetite (Metabolism and nutrition disorders) | 22 (25)
Irritability (Psychiatric disorders) | 38 (50)
Somnolence (Nervous system disorders) | 25 (30)
Crying (General disorders) | 28 (35)
Injection Site Bruising (General disorders) | 9 (10)
Injection Site Erythema (General disorders) | 25 (31)
Injection Site Induration (General disorders) | 12 (12)
Injection Site Pain (General disorders) | 44 (53)
Injection Site Swelling (General disorders) | 12 (14)
Pyrexia (General disorders) | 9 (11)

LIMITATIONS AND CAVEATS:
The main efficacy cohort was not conducted due to shift in the global influenza vaccine guidelines. Hence, no analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04544267/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04544267/SAP_001.pdf